CLINICAL TRIAL: NCT03907670
Title: Clinical and Immunological Outcome in Chronic Myloid Leukemic Patients Treated With Tyrosine Kinase Inhibitor: Assuit University Hospitals Insight
Brief Title: Chronic Myloid Leukemic Patients Treated With Tyrosine Kinase Inhibitor
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Esraa Nageh Adam, principal investigator, Assiut University
Other Study IDs: EAdam
Record Dates: First submitted 2019-04-05; First posted 2019-04-09 (Actual); Last update posted 2019-09-30 (Actual); Status verified 2019-04

CONDITIONS: Chronic Phase Chronic Myelogenous Leukemia
Keywords: chronic myeloid leukemia; Tyrosine kinase inhibitors
MeSH Terms: conditions — Leukemia, Myeloid, Chronic-Phase; Leukemia, Myelogenous, Chronic, BCR-ABL Positive

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- CML patients who will receive imatinib: Patients with chronic myeloid leukemia newly diagnosed, who will receive Tyrosine Kinase inhibitor treatment (imatinib)measure the fluctuations in the levels of sCTLA-4, TGFβ1, and PDMPs, and to clarify the clinical significance of these biomarkers during TKI therapy in patients with CML
- CML patients who will receive nilotinib: Patients with chronic myeloid leukemia newly diagnosed, who will receive Tyrosine Kinase inhibitor treatment(nilotinib)measure the fluctuations in the levels of sCTLA-4, TGFβ1, and PDMPs, and to clarify the clinical significance of these biomarkers during TKI therapy in patients with CML
- CML patients who will receive dasatinib: Patients with chronic myeloid leukemia newly diagnosed, who will receive Tyrosine Kinase inhibitor treatment(dasatinib) measure the fluctuations in the levels of sCTLA-4, TGFβ1, and PDMPs, and to clarify the clinical significance of these biomarkers during TKI therapy in patients with CML

SUMMARY:
The aim of the study is to assesse the levels of various biomarkers, specifically interleukin (IL)-6, platelet-derived microparticles (PDMPs), 11, 12 soluble vascular cell adhesion molecule 1 (sVCAM-1), transforming growth factor (TGF) β1, and sCTLA-4, in TKI-treated patients with CML.

To measure the fluctuations in the levels of sCTLA-4, TGFβ1, and PDMPs, and to clarify the clinical significance of these biomarkers during TKI therapy in patients with CML..

DETAILED DESCRIPTION:
Chronic myelogenous leukemia (CML) is a myeloproliferative disorder in which leukemic cells display the Philadelphia chromosome generated from a reciprocal t(9:22) (q34:q11) translocation.1 The chromosome 9 and chromosome 22 transposal of t (9:22) and (q34:q11) causes the cancer gene C-ABL at 9q34 to link with the BCR gene at 22q11, forming the BCR-ABL gene on chromosome 22.2 CML is presented by constitutional complaints (fatigue, weight loss, and fever), those related to splenomegaly (abdominal fullness, anorexia, abdominal pain, and early satiety) and bleeding tendency (easy bruising or bleeding) are most frequent symptoms. Splenomegaly (≥ 95%), sternal tenderness, hepatomegaly, purpura, and retinal hemorrhage are commonly reported signs at physical exam. To diagnose CML, doctors use a variety of tests to analyze the blood and marrow cells.

*Complete Blood Count (CBC). This test is used to measure the number and types of cells in the blood. People with CML often have:

* Decreased hemoglobin concentration
* Increased white blood cell count, often to very high levels
* Possible increase or decrease in the number of platelets depending on the severity

Blood cells are stained (dyed) and examined with a light microscope. These samples show:

* Specific pattern of white blood cells
* Small proportion of immature cells (leukemic blast cells and promyelocytes)
* Larger proportion of maturing and fully matured white blood cells (myelocytes and neutrophils).

These blast cells, promyelocytes and myelocytes are normally not present in the blood of healthy individuals

* Bone Marrow Aspiration and Biopsy.
* Cytogenetic Analysis.
* FISH (Fluorescence In Situ Hybridization).
* Polymerase Chain Reaction (PCR).

The disease is classically staged into chronic phase (CP, most patients at presentation), accelerated phase (AP) and blast phase (BP).3 Many definitions have been used for these stages, but all the data generated from the tyrosine kinase inhibitor (TKI) studies has used the historically standard definition where AP is defined by the presence of one or more of the following: ≥15% blasts in the peripheral blood or bone marrow, ≥20% basophils in the peripheral blood , platelets <100,000/μL unrelated to treatment or the development of cytogenetic evolution. Blast phase is defined by the presence of ≥30% blasts in the peripheral blood or bone marrow, the presence of clusters of blasts in marrow or the presence of extramedullary disease with immature cells (i.e., a myeloid sarcoma).4 Progression to BP occurs at a median of 3-5 years from diagnosis in untreated patients, with or without an intervening identifiable AP.5. After initiating therapy for CML, patients should be monitored for treatment response assessment. The process of monitoring response to therapy is important to determine if an adequate response is being achieved, or if patients should be transitioned to a higher dose or different therapy Since therapy is continued indefinitely and relapse occurs upon cessation of therapy in most patients, it is critical that the disease is closely monitored. Continued monitoring over time is needed, even in the setting of an optimal response, in order to detect and treat potential recurrence. Specific response criteria, including optimal, suboptimal, and failure have been established to guide appropriate increase or change of therapy

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed CML patients
2. Receive TKI treatment (imatinib, nilotinib, dasatinib) selected among those admitted to the investigator's hospital.
3. Ageing group 20yr up to 80 yr.

Exclusion Criteria:

1. CML patients who previously treated with TKI.
2. Age below 20 yrs.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 45 patients with chronic myeloid leukemia newly diagnosed, who will receive TKI treatment (imatinib, nilotinib, dasatinib
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2019-10-01 (Estimated); Primary Completion 2020-10-01 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
assessment of CML patients receiving tyrosine kinase inhibitors | 6 months
  Assesse the levels of various biomarkers, especifically 1-interleukin (IL)-6, 2- platelet-derived microparticles (PDMPs),3- 17-20 soluble vascular cell adhesion molecule 1(sVCAM-1),4- Transforming growth factor (TGF) β1, and sCTLA-4, in TKI-treated patients with CML